CLINICAL TRIAL: NCT02480569
Title: Trial to Compare FFR Measurement With a Non-Side-Hole Guide Catheter Vs. a Side-Hole Guide Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Emmanouil S Brilakis, MD, PhD, North Texas Veterans Healthcare System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-033
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Side-Hole Catheter (Experimental): 2 FFR measurements from an engaged side-hole guide catheter and a disengaged side-hole guide catheter
  Interventions: Other: FFR Measurement
- Non-Side-Hole Catheter (Experimental): 2 FFR measurements from an engaged non-side-hole guide catheter and a disengaged non-side-hole guide catheter
  Interventions: Other: FFR Measurement

INTERVENTIONS:
Other: FFR Measurement

SUMMARY:
The investigators propose a single center prospective study that will assess two different strategies for measuring Fractional Flow Reserve (FFR) in patients undergoing clinically-indicated coronary angiography in whom FFR measurement is indicated. FFR will be measured with a non-side hole guide catheter (with the guide catheter both engaged and disengaged from the coronary ostium) and with a side-hole guide catheter (with the guide catheter both engaged and disengaged from the coronary ostium) to determine, whether measurements obtained with an engaged side-hole guide catheter are more accurate as compared with those obtained with the engaged non-side hole catheter.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a clinically indicated coronary catheterization
* Need FFR of a coronary artery lesion
* Agree to participate and able to provide informed consent

Exclusion Criteria:

* Significant difficulty advancing the pressure measuring guidewire into the coronary artery
* Severe chronic obstructive pulmonary disease
* Severe ostial disease (>70% diameter stenosis within 5 mm from the coronary artery ostium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
FFR measurement using a guide catheter with and without side holes | Less than 1 hour during the coronary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States